CLINICAL TRIAL: NCT03116815
Title: The Feasibility of a Web-based Application to Monitor Home Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Holly J. Mattix-Kramer, Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 209116
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: blood pressure; monitoring; hypertension; patient reported outcomes
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This single arm study will examine use of the MyChart web-application whereby patients directly record their home blood pressure readings into their electronic health record with this web-based application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Intervention is the use of the MyChart web-application whereby participants record their home blood pressure readings directly into their electronic medical record. Their physicians are then alerted of these blood pressure readings.
  Interventions: Other: Direct input of home blood pressure readings via MyChart

INTERVENTIONS:
Other: Direct input of home blood pressure readings via MyChart — Participants will record home blood pressure readings directly into the electronic health record via the MyChart application

SUMMARY:
Control of hypertension remains one of the most important interventions available to clinicians to reduce risk of cardiovascular disease, kidney disease and stroke. Self-measured home blood pressure monitoring plus additional support has been shown to reduce blood pressure in adults with previously uncontrolled hypertension. Most previous studies have utilized healthcare personnel to facilitate communication of home blood pressure levels to physicians and did not provide methods to directly transmit self-measured blood home blood pressure levels to physicians via the electronic health record. Emerging technology now provides the ability for patient's to upload self-measured blood pressure levels into their own medical record which may eliminate the need for additional health personnel. This study will examine the feasibility, patient adherence and physician and patient perceptions of a web-based application which will facilitate direct input of self-measured home blood pressure levels and patient reported symptoms directly into the electronic health record with message alerts to the provider for hypertension management. Up to 10 Loyola primary care physicians and 20 of their respective patients age 50 years and older who have a smart phone device or home computer and have treated hypertension will be enrolled. The study will utilize the existing web-application called MyChart. MyChart is the name of the web-based application and it is not an acronym. Enrolled patients will download the existing MyChart web-based application on their smart phone device or home computer and will record home blood pressure measurements using their home blood pressure machine into their smart phone application. The MyChart application is available to all patients receiving care in the Loyola Health Care System. The blood pressure readings and patient reported symptoms will then be available for their physicians to review within the electronic health record. After using the web-based application for two months, both patients and physicians will be asked to participate in focus groups and interviews, respectively, to determine their perceptions and satisfaction with the web-based application. Data from this feasibility study may be used to guide a future clinical trial of hypertension management that examines the effectiveness of the MyChart web-based application for frequent blood pressure monitoring compared to standard care.

DETAILED DESCRIPTION:
Observational studies and clinical trials have demonstrated that clinicians fail to intensify therapy in hypertensive management despite patients not meeting goal. For this reason, patient centered tools can help facilitate meeting goals with the provider. Web-based communication combined with provider care management successfully lowered blood pressure to <140/90 mm Hg in prior studies of patients with hypertension. Emerging technology now provides the ability for patients to upload self-measured home blood pressure information into their own medical record which may eliminate the need for additional health personnel. This study will investigate the feasibility of health informatics to facilitate better compliance and safety for both provider and patient for hypertension management. The home blood pressure readings along with patient reported symptoms will be recorded using the MyChart, a web-based tool available to all patients receiving care at Loyola University Medical Center. MyChart can be accessed with a hand-held device or home computer. After enrollment, patients will receive a notice every two weeks via MyChart to upload home blood pressure values and patient reported symptoms. This information entered into MyChart by patients will be placed into the electronic health record in a home vital signs flow sheet, which will be separate from the flow sheet of vital signs measured in the clinic. Physicians will receive an alert message when patients upload the blood pressure data. The alert message will provide physicians with the average blood pressure value over the two weeks and will provide simple guidance on whether actions, such as titrating existing medication should be taken (based on whether BP is ≥ 140/90 mmHg). Patients will also be able to track their own home blood pressure values using the MyChart application. As a first step, we are first examining the feasibility of this web-based application and determining the perceptions of both patients and physicians.

ELIGIBILITY:
* Inclusion Criteria:

  * Willing to participate in all study procedures
  * Potential subject owns a personal device and is able to run the web-application
  * Physician directed blood pressure goal is < 140/90 mmHg
* Exclusion Criteria:

  * No use of blood pressure lowering medications
  * Arm circumference too large or small to allow accurate blood pressure measurement
  * A medical condition likely to limit survival to less than 6 months, or a cancer diagnosed and treated within the past two years that, in the judgment of clinical study staff, would compromise a participant's ability to complete the study
  * Inability to give informed consent
  * History of systolic heart failure (ejection fraction < 35%)
  * History of stroke
  * History of proteinuria ≥ 1 gram in a 24 hour urine collection or a random urine albumin/creatinine ratio ≥ 300 mg/g or a random urine protein/creatinine ratio ≥ 300 mg/g

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
The total number of patients screened for the study | 30 days
  The total number of patients who were examined for study eligibility
The total number of patients who meet study eligibility | 30 days
  The total number of patients who are screened for the study and meet study eligibility
The total number of patients who provide written informed consent to participate in the study | 30 days
  The total number of patients who enroll in the study and provide written informed consent
The number of home blood pressure readings submitted by patients to the MyChart web-based application | 60 days
  The actual number of home blood pressure readings that are recorded in the electronic health record as submitted via MyChart
Change in systolic blood pressure | 60 days
  Change in systolic blood pressure
Change in diastolic blood pressure | 60 days
  Change in diastolic blood pressure
Physician actions based on home blood pressure readings | 60 days
  Total number of times a physician escalates or de-escalates blood pressure lowering medications for a study participant
Correlation between office and home blood pressure readings | one day
  Correlation between the office blood pressure measurement using the clinic Omron machine and the patient's home blood pressure cuff
Adverse events | 60 days
  Total number of patient reported adverse events and all hospitalizations and emergency room visits
Patient reported outcomes | 60 days
  The percentage quality of life questionnaires completed by the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Holly Kramer, MD MPH, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No